CLINICAL TRIAL: NCT06929260
Title: A Phase I, Open-label, Fixed-sequence Study to Evaluate the Effect of Ceralasertib on Pharmacokinetics of Drug X, Drug Y and Drug Z in Participants With Advanced Solid Tumours
Brief Title: A Study to Evaluate the Effect of Ceralasertib on Drug X, Drug Y and Drug Z
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study terminated because the clinical development programme for Ceralasertib has been discontinued.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D533BC00003; 2024-516611-24-00 (Other: EU CT Number)
Record Dates: First submitted 2025-04-14; First posted 2025-04-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumours
Keywords: Pharmacokinetics; Drug-drug interactions
MeSH Terms: interventions — ceralasertib; factor IX, factor VII, factor X, prothrombin drug combination; drug XX Z

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ceralasertib, Drug X, Drug Y and Drug Z (Experimental): Participants will receive ceralasertib twice daily (BD) from Day 1 to Day 7. Participants will also receive a single dose of Drug X on Day 5 and Day 22. Similarly, a single dose of Drug Y and Drug Z on Day 7 and Day 28.
  Interventions: Drug: Ceralasertib; Drug: Drug X; Drug: Drug Y; Drug: Drug Z

INTERVENTIONS:
Drug: Ceralasertib — Participants will receive repeated dosing of ceralasertib from Day 1 to Day 7 until steady state.
  Other Names: AZD6738
Drug: Drug X — Participants will receive a single dose of Drug X on Day 5 and Day 22.
Drug: Drug Y — Participants will receive a single dose of Drug Y on Day 7 and Day 28.
Drug: Drug Z — Participants will receive a single dose of Drug Z on Day 7 and Day 28.

SUMMARY:
The study aims to assess the effect of ceralasertib on the pharmacokinetics (PK) of Drug X, Drug Y and Drug Z in participants with advanced solid tumours.

DETAILED DESCRIPTION:
This is an open-label, 3-period fixed-sequence study. The study will comprise of -

* Screening Visit (Visit 1)
* Period 1 (Visit 2)
* Period 2 (Visit 3)
* Period 3 (Visit 4)
* Follow-up Visit (Visit 5)

A wash-out period of no less than 48 hours in each period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic solid tumour(s) of non-small cell lung cancer, ovarian cancer, endometrial cancer, breast cancer or prostate cancer at Screening.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 with no deterioration over the 2 weeks prior to dosing.
* Ability to swallow and retain oral medication.
* Minimum life expectancy ≥ 12 weeks in the opinion of the Investigator.
* Adequate organ and marrow function during Screening.
* Body weight > 30 kg and no cancer-associated cachexia.
* Contraceptive use by participants or participant partners should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Diagnosis of ataxia telangiectasia (ATR).
* History of another primary malignancy except for:

  1. Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of the study intervention and of low potential risk for recurrence.
  2. Basal cell carcinoma of the skin.
  3. Curatively treated in situ cancer of the cervix.
  4. Ductal carcinoma in situ.
  5. Curatively treated lymphomas (without bone marrow involvement).
  6. Squamous cell carcinoma of the skin or lentigo maligna that has undergone potentially curative therapy.
  7. Adequately treated carcinoma in situ without evidence of disease.
* History of leptomeningeal carcinomatosis.
* History of myelodysplastic syndromes (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML (as determined by prior diagnostic investigation).
* Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study intervention.
* Spinal cord compression or brain metastases for at least 4 weeks prior to start of study intervention unless asymptomatic and stable.
* Persistent toxicities, with the exception of alopecia and vitiligo, caused by previous anti-cancer therapy.
* Participants with any known predisposition to bleeding.
* Refractory nausea and vomiting, chronic gastrointestinal diseases associated with diarrhoea, or previous significant bowel resection, with clinically significant sequelae that would preclude adequate absorption of ceralasertib.
* Any of the following cardiac criteria or cardiovascular diseases -

  1. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG.
  2. Any factors that increase the risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age.
  3. Participants at risk of brain perfusion problems.
  4. Participants with relative hypotension or uncontrolled hypertension requiring clinical intervention.
  5. Hypertensive heart disease with significant left ventricular hypertrophy or clinically significant valvular heart disease.
  6. History of atrial or ventricular arrhythmia requiring treatment.
  7. Transient ischaemic attack or stroke within 6 months prior to Screening.
* Any participant with active infection requiring systemic antibiotics, antifungal or antiviral drugs.
* Participants with confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or active infection requiring systemic antibiotics, antifungal or antiviral drugs.
* Any prior treatment with an ATR inhibitor or checkpoint kinase inhibitor.
* Any concomitant treatment of central nervous system depressants, opioids, and centrally acting anti-hypertensive agents.
* Receipt of the last dose anti-cancer therapy within 4 weeks or 5 half-lives prior to the first dose of ceralasertib, whichever is shorter.
* Concomitant use of proton pump inhibitors, histamine H2 receptor antagonists, and other anti-acid agents.
* Palliative radiotherapy with a limited field of radiation within 2 weeks.
* Receiving or intend to receive any prescription or non-prescription drugs within 7 days or 5 half-lives before first dose of study intervention.
* Use of tobacco- or nicotine-containing products within 3 months prior to check-in or history of drug or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) | From Day 5 to Day 30
  To assess the effect of ceralasertib on the PK of Drug X, Drug Y and Drug Z.
Area under plasma concentration-time curve from time 0 to last quantifiable concentration (AUClast) | From Day 5 to Day 30
  To assess the effect of ceralasertib on the PK of Drug X, Drug Y and Drug Z.
Maximum observed concentration (Cmax) | From Day 5 to Day 30
  To assess the effect of ceralasertib on the PK of Drug X, Drug Y and Drug Z.
Plasma terminal elimination half-life (plasma t1/2λz) | From Day 5 to Day 30
  To assess the effect of ceralasertib on the PK of Drug X, Drug Y and Drug Z.
Terminal elimination rate constante (λz) | From Day 5 to Day 30
  To assess the effect of ceralasertib on the PK of Drug X, Drug Y and Drug Z.
Time to Reach Maximum Concentration Following Drug Administration (tmax) | From Day 5 to Day 30
  To assess the effect of ceralasertib on the PK of Drug X, Drug Y and Drug Z.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From Screening to follow up visit, for up to 65 days
  To assess the safety and tolerability of ceralasertib.
Trough concentrations of ceralasertib. | Day 4 to Day 7
  To assess ceralasertib steady state.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST /Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/